CLINICAL TRIAL: NCT02780960
Title: HPV Self-sampling as a Test of Cure After Treatment of Cervical Intra-epithelial Neoplasia
Brief Title: Human Papillomavirus (HPV) Self-sampling as a Test of Cure After Treatment of Cervical Intra-epithelial Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Manuela Viviano, Dr, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-285
Record Dates: First submitted 2016-05-13; First posted 2016-05-24 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Cervical Intra-epithelial Neoplasia Grade 1 or Worse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HPV self-testing (Experimental): Patients will perform HPV self-testing at home, prior to their follow-up visit. At the colposcopy visit, the doctor or nurse will also perform HPV testing. This procedure will be repeated at 6 and 12 months following LEEP.
  Interventions: Device: HPV self-testing

INTERVENTIONS:
Device: HPV self-testing — Patients will perform HPV testing themselves at home.

SUMMARY:
The purpose of this study is to evaluate the performance of HPV self-sampling (self-HPV) in detecting residual/recurrent disease in women treated by loop electro-surgical excision (LEEP) for CIN1+.

DETAILED DESCRIPTION:
The HPV test is an efficient method to assess the long-term risk of residual/recurrent disease in women treated for cervical intraepithelial neoplasia grade 1 or worse (CIN1+).

Women treated by LEEP for CIN1+ will be invited to participate. Follow-up visits will be performed at 6 months and 12 months after treatment and will include cytology, colposcopy when indicated and HPV testing. Two weeks before each follow-up visit at the colposcopy clinic, a home-based Self-HPV will be organized. A sample of 168 women will be included. Agreement between the two methods (Dr-HPV vs. S-HPV) will be measured using the kappa statistic (κ).

the investigators expect to find that Self-HPV may be an accurate method to predict residual and recurrent disease in women previously treated by LEEP.

ELIGIBILITY:
Inclusion Criteria:

* attending colposcopy clinic
* biopsy-proven CIN1+ lesion
* understands study procedures and accepts voluntarily to participate by signing the informed consent form

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-05; Primary Completion 2020-09 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with CIN | 12 months
  Number of patients with CIN after LEEP.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Derived] Viviano M, Vassilakos P, Meyer-Hamme U, Grangier L, Emery SL, Malinverno MU, Petignat P. HPV self-sampling in the follow-up of women after treatment of cervical intra-epithelial neoplasia: A prospective study in a high-income country. Prev Med Rep. 2021 Sep 20;24:101564. doi: 10.1016/j.pmedr.2021.101564. eCollection 2021 Dec. PMID 34976630